CLINICAL TRIAL: NCT02493426
Title: Single Dose Intranasal Oxytocin (IN-OT) Versus Placebo in Autism: Examining Cognitive Effects
Brief Title: Single Dose Intranasal Oxytocin and Cognitive Effects in Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: PSYCH-2016-21943
Record Dates: First submitted 2015-07-06; First posted 2015-07-09 (Estimated); Results first posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Saline Nasal spray designed to look and feel like the drug intervention
  Interventions: Drug: Placebo
- Intranasal Oxytocin (Experimental): Oxytocin nasal spray designed to look as seem exactly like Placebo
  Interventions: Drug: Intranasal Oxytocin

INTERVENTIONS:
Drug: Intranasal Oxytocin
  Arms: Intranasal Oxytocin
Drug: Placebo
  Arms: Placebo

SUMMARY:
Autism spectrum disorder (ASD) is a group of severe, life-long developmental disorders. Oxytocin (OT) is a neurohormone involved in both repetitive/rigid and social behaviors. This study is focusing on how a single dose of intranasal OT (IN-OT) affects cognitive rigidity and social perception tasks. Taking OT as a spray through the nose increases social and decreases repetitive behavior in some adults with ASD, and we are exploring if it helps children with ASD similarly. However, it is unclear whether every person with ASD has an abnormal OT level, and if OT affects restrictive or social behavior differently. Consequently, we aim to study whether OT treatment can be effective in treating subgroups with specific features of ASD. We will use approaches utilizing both behavioral and physiological responses to clarify the role of OT in ASD. We will develop a deeper understanding of the range of social and rigid behaviors and use that information to identify persons with ASD who would benefit from OT treatment. Potential subjects will be asked if they want to participate in two sessions in our clinical laboratory where they will get either single dose IN-OT or placebo. After receiving the substance, they will be asked to do a handful of tasks while we monitor heart rate, eye movements, and collect baseline and post intranasal blood, urine and saliva. The levels of hormones, metabolites and peptides related to or interacting with OT will be measures in the collected samples of blood plasma, urine and saliva. Additionally DNA will be extracted from the blood samples to study genes related to OT and ASD.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be between 5 and 40 years of age.
* All subjects will have a diagnosis of autistic disorder or ASD that was confirmed by administration of the Autism Diagnostic Observation Schedule-WPS (ADOS-WPS) (30).
* Eligible participants must be able to perform the cognitive learning tasks.

Exclusion Criteria:

* Although we acknowledge that concomitant medications, or other types of intervention, may potentially bias study results, participants will be allowed to stay on concomitant medications and non-pharmacologic treatments, provided that no changes are made within 3 months prior to baseline and that no changes are made during the study.
* Individuals that are on antipsychotic drugs will be excluded from participation. All subjects must lack a significant medical history.
* Subjects with any condition, including alcohol and drug abuse, which might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being will be excluded.
* This includes, but is not limited to impairment of renal function, evidence or history of malignancy or any significant hematological, endocrine, respiratory, hepatic, cardiovascular or gastrointestinal disease.
* All female subjects of childbearing capacity will have a urine pregnancy test (a positive test will exclude the subject from participation).
* A pregnancy test will be conducted at both visits prior to drug administration. Uterine contractions may occur in women and are more likely to occur in pregnant women, especially towards the end of pregnancy.
* As a result, we exclude pregnant female patients, sexually active female patients on hormonal birth control and sexually active females who do not use two types of non-hormonal birth control.
* All interested potential subjects will be contacted via phone. If they meet eligibility criteria, two sessions that are approximately two weeks apart and approximately the same time of day will be scheduled. At their first visit, we will review the study and undergo informed consent procedures. Overall study procedures per visit are estimated to take approximately 2-3 hours per session, and are detailed in Table 2.

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suma Jacob, MD/PhD, Principal Investigator — University of Minnesota
Locations (1):
- Center for Neurobehavioral Development, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then Intranasal Oxytocin: Saline Nasal spray designed to look and feel like the drug intervention
  Placebo
- Intranasal Oxytocin Then Placebo: Oxytocin nasal spray designed to look as seem exactly like Placebo
  Intranasal Oxytocin
Period: Overall Study
Arm/Group | Placebo Then Intranasal Oxytocin | Intranasal Oxytocin Then Placebo
Started | 14 | 13
Completed | 14 | 12
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants (cross-over design)
Arm/Group | All Participants
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 19
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Reading the Mind in the Eyes Task (RMET)
Description: Social Cognition Task-- We are reporting raw score (# of correct responses) Minimum value is 0 and maximum value is 28. A higher score means better performance / outcome.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: total raw score
Groups:
- Placebo Then Oxytocin: Saline Nasal spray designed to look and feel like the drug intervention
  Placebo
Arm/Group | Placebo Then Oxytocin | Intranasal Oxytocin Then Placebo
Number analyzed (Participants) | 14 | 12
total raw score
  Intervention Period 1 | 18.07 (4.48) | 18.08 (2.47)
  Intervention Period 2 | 17.86 (4.77) | 18.09 (3.08)

2. Primary Outcome: Rapid Automatized Naming (RAN)
Description: Cognitive Rigidity Task for >10 years old-- Time to name attribute of stimulus requested; minimum time is 0, there is no maximum time. Lower score is better.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: naming time (seconds)
Arm/Group | Placebo Then Oxytocin | Intranasal Oxytocin Then Placebo
Number analyzed (Participants) | 10 | 8
naming time (seconds)
  Symbolic: Intervention Period 1 | 18.08 (4.69) | 16.13 (6.21)
  Symbolic: Intervention Period 2 | 17.98 (5.71) | 15.28 (4.63)
  Non-symbolic: Intervention Period 1 | 27.93 (6.02) | 24.13 (6.31)
  Non-symbolic: Intervention Period 2 | 28.70 (6.95) | 23.31 (7.16)

3. Primary Outcome: Dynamic Affect Recognition Evaluation (DARE)
Description: Task Performance with Physiological Data. We reported the raw score - total number correct. Minimum is 0, maximum is 12. Higher score means better performance / outcome.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: total raw score
Arm/Group | Placebo Then Oxytocin | Intranasal Oxytocin Then Placebo
Number analyzed (Participants) | 14 | 12
total raw score
  Intervention Period 1 | 8.5 (3.32) | 8.45 (3.67)
  Intervention Period 2 | 8.36 (3.43) | 8.92 (4.01)

ADVERSE EVENTS:
Time Frame: 6 weeks per participant
Groups:
- Placebo: Saline Nasal spray designed to look and feel like the drug intervention, then Placebo
- Intranasal Oxytocin: Oxytocin nasal spray designed to look as seem exactly like Placebo, then Intranasal Oxytocin
Arm/Group | Placebo | Intranasal Oxytocin
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 14/27 | 13/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=27) | Intranasal Oxytocin (N=27)
Headache (General disorders) | 0 (0) | 1 (1)
Bloody nose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Mouth pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Greater awakeness (General disorders) | 0 (0) | 1 (1)
Energized (General disorders) | 0 (0) | 1 (1)
Lightheadedness (General disorders) | 1 (1) | 1 (1)
Greater calmness (Nervous system disorders) | 4 (4) | 2 (2)
Less anxiety (Nervous system disorders) | 3 (3) | 1 (1)
Perseveration (Nervous system disorders) | 1 (1) | 0 (0)
Less flexibility (General disorders) | 1 (1) | 1 (1)
Loss of appetite (General disorders) | 1 (1) | 1 (1)
Agitation (Nervous system disorders) | 0 (0) | 1 (1)
Drowsiness (Nervous system disorders) | 1 (1) | 0 (0)
Dry mouth (General disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chill (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-06-25): https://cdn.clinicaltrials.gov/large-docs/26/NCT02493426/Prot_SAP_000.pdf
  • Informed Consent Form (2015-07-16): https://cdn.clinicaltrials.gov/large-docs/26/NCT02493426/ICF_001.pdf